CLINICAL TRIAL: NCT00667498
Title: Metabolic Effect of Metformin in Obese Insulin Resistant Adolescents With Normal Glucose Tolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Tania S. Burgert, M.D., Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0311026134
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Pediatric Obesity; Insulin Resistance; Hyperinsulinemia
Keywords: Pediatric Obesity; Insulin Resistance; Hyperinsulinemia; Metformin; Glucose Tolerance; Microalbuminuria; Adolescents; Visceral Fat
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Hyperinsulinism | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Metformin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — The subject will receive either metformin or placebo drug, given as 500mg tablets (or corresponding placebos) necessary to increase the dose incrementally over a three week period.
  The time it takes to incrementally increase the dose to the desired dose of 500mg in am and 1000mg in pm will count as intervention time. Both the metformin and placebo group will also be given a multivitamin with vitamin B12 to avoid potential anemia.
  Other Names: Glucophage, Glucophage XR, Glumetza, Fortamet, Riomet
  Arms: 1
Drug: Placebo — The subject will receive either metformin or placebo drug, given as 500mg tablets (or corresponding placebos) necessary to increase the dose incrementally over a three week period.
  The time it takes to incrementally increase the dose to the desired dose of 500mg in am and 1000mg in pm will count as intervention time. Both the metformin and placebo group will also be given a multivitamin with vitamin B12 to avoid potential anemia.
  Arms: 2

SUMMARY:
The primary objective of this randomized, parallel group, double-blind, placebo-controlled study is to determine whether treatment with metformin enhances insulin sensitivity in a group of ethnically diverse obese insulin-resistant adolescents with normal glucose tolerance.

DETAILED DESCRIPTION:
First Visit

Patients who agree to participate in this research study, will have an initial screening where the subject will be asked about his/her health, a sample of blood will be drawn, the subject will be examined, and an oral glucose tolerance (OGTT) test will be done.

* OGTT: The study takes about four hours and will begin on an "empty stomach." A small I.V. will be placed in a vein in the subject's arm. The I.V. will allow a member of the research team to take small amounts of blood for measuring glucose and other substances that circulate in the blood. About 7 tablespoons of blood will be drawn in total during the OGTT. The I.V. will remain in place all during the study. At the beginning of the study, the subject will be asked to drink about 8 ounces (one cup) of a high sugar cola- or orange-flavored drink.

If the subject meets all the requirements to be in the study and has a normal glucose tolerance test, he/she will be randomized to either the intensely (Euglycemic hyperinsulinemic clamp) or standard studied group and have the following six or seven tests performed: DEXA scan and Tanita, exercise step test, PAT test, MRI (Abdominal scan), MRS (leg scan), and Euglycemic hyperinsulinemic clamp (intensely studied group only). All of the tests are described below. Females will have a urine pregnancy test before each of these tests. If positive, the subject will not be allowed to participate/continue with the study.

* DEXA / Tanita: The DEXA scan will measure how much muscle and fat is in the subject's body and how dense the subject's bones are using an x-ray technique. Directly after the DEXA Scan, the subject's percentage of body fat will be measured using a Tanita scale.
* Exercise Step Test: The subject will be asked to step up and down two steps 20 times at their own pace. We will measure the subject's heart rate directly before and for three minutes after this exercise. After a ten minute break, the test will be repeated.
* Peripheral Arterial Tonometry (PAT): This test will allow us to evaluate the response of the small blood vessels in the subject's arm to changes in nerve signals to them. During this test, we will put a probe (similar to a tight-fitting glove) on one finger of each of the subject's hands and take some measurements for about five minutes. The probes contain latex, so this test will not be performed on subjects who are allergic to latex. Following these measurements, we will block blood flow to one of the hands for five minutes by putting a blood pressure cuff on one of the arms and inflating the cuff. After the pressure in the cuff is released, we will take more measurements for about five minutes.
* MRI (Belly Scan): Magnetic Resonance Imaging (MRI) will be used to take pictures of the subject's belly. These pictures will allow us to calculate how much fat the subject has just below the skin and how much fat is deeper inside the belly. We will also be able to estimate the percentage of fat in the subject's liver.
* MRS (Leg scan): We will measure how much fat is in the subject's calf muscle using magnetic resonance spectroscopy (MRS).
* Insulin, Glucose and Glycerol Infusion Study (Euglycemic hyperinsulinemic clamp): A small I.V. will be placed into a vein in each arm. One I.V. will be used to take out small amounts of blood for measuring the blood sugar and other substances that circulate in the blood. The other I.V. will be used to infuse insulin, glucose, and glycerol into the subject's blood. Insulin is a hormone that helps bring blood sugar into the cells. Glycerol is a component of fat that is normally present in a person's body.

This infusion will not affect the subject's blood sugar in a harmful manner. It will allow us to follow the release of glucose from the liver and glycerol from fat tissue.

The subject's blood sugar will be checked closely during the study by taking blood samples from the second I.V. Readings of the blood sugar on each sample will be made at the bedside. If the blood sugar starts to fall, it can be fixed right away. At the end of another three hours, the infusion will be stopped and the subject will eat a meal that will be provided for him/her. The infusion of glucose will be reduced while the subject is eating until the subject's blood sugar is stable. This test takes about 6 hours. The total amount of blood drawn during this test will be less than 8 tablespoons or about half a cup.

Indirect calorimetry is a way to measure how much sugar and fat a person is burning when we give insulin. Testing how much fat and sugar a subject burns is an important part of the insulin, glucose, and glycerol infusion study. Therefore we will ask the subject to wear a plastic hood (like an astronaut space helmet) before starting the infusion of insulin and at two other times during the study.

Taking Metformin or Placebo

Once the subject has completed the six (standard studied group) or seven (intensely studied group only) tests described above, as well as two urine tests for protein, he/she will be randomized to either:

* Take Metformin; or
* Take a placebo pill

The subject will begin by taking one pill (either Metformin or placebo) every day, just before supper. The dose will be slowly increased as follows:

Week 1: Before breakfast = 0 and Before supper = 1 (500mg); Week 2: Before breakfast = 1 (500mg) and Before supper = 1 (500mg); Week 3-14: Before breakfast = 1 (500mg) and Before supper = 2 (500mg)

The subject will be taking the pills for 3 1/2 months, during which time we will ask that he/she keep a diary of any complaints, problems, or symptoms. Neither the subject, the subject's doctor, nor any of the members of the research team will find out which pill the subject was taking until the end of the study.

Monthly Follow-up

Subjects will be asked to come back every month for a physical exam. We will measure their height, weight, and blood pressure each time. A urine pregnancy test will be done on all female participants at every visit. At the subject's first follow up visit we will draw a small amount of blood and run tests to make sure the subject is healthy. We will ask the subject and his/her parent about any symptoms that the subject has had, any pills that he/she might have missed taking, and the use of other medications. We will measure the subject's vitamin B12 level on his/her third follow up visit.

End of Study

About three months after the subject begins taking the Metformin or placebo pills, he/she will repeat the tests described above (oral glucose tolerance test, DEXA and Tanita, exercise step test, PAT test, MRI, and MRS). In the sub-group of participants who had the glucose, insulin, and glycerol infusion test, this will also be repeated at the end of the study.

Open Label Phase (Taking Metformin)

After the tests described above are completed, all participants (even if they had been assigned a placebo pill) will be given the choice of taking Metformin for the next six months. If the subject does choose to continue, we will continue to monitor him/her monthly, as described in the section above on monthly follow-up. At the end of the additional six months, we will repeat all the tests that the subject had at the beginning of the study. For the intensely studied group, this includes the insulin, glucose and glycerol infusion.

ELIGIBILITY:
Inclusion Criteria:

* Attending weight management clinic at Yale New Haven Hospital
* Good general health, taking no other medication on a chronic basis
* Age 13 to 17 yrs in puberty (girls: breast Tanner stage II to IV, and boys: testes size > 6 ml)
* The presence of insulin resistance, defined by fasting insulin levels greater than 30 µU/ml, and HOMA insulin resistance index > 6
* Normal glucose tolerance based on a 2-hr plasma glucose (<140 mg/dl) after the OGTT.
* All female subjects must have a negative urine pregnancy test during the study visits and must use an effective method of contraception if they are sexually active. Without their parent(s) present, all potential female subjects will be asked about their sexual activity and the specific form of contraception they are using.

Exclusion Criteria:

* Baseline creatinine > 1.0 mg/dl
* Hepatic disease with elevated liver function test (ALT or AST) ≥ 2 X the upper limits of normal
* Pregnancy
* Presence of other endocrinopathies; except treated hypothyroidism on stable replacement doses of thyroid hormone
* Presence of cardiac, pulmonary or other significant chronic illness
* Adolescents with psychiatric disorder, claustrophobia or with substance abuse
* Recent use (within six months) of anorexic agents
* Presence of anemia (hematocrit < 35)
* Mixed ethnic background (defined as two parents of different ethnicity)
* Adolescents with metal implants (i.e. cardiac pace maker, metal prostheses, bullet remnants)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Assessment of insulin sensitivity: Whole Body Insulin Sensitivity Index (WBISI), Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), and Euglycemic hyperinsulinemic clamp | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Waist to hip circumference ratio | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Muscle lipid content | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Total body fat | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Abdominal fat mass | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Hepatic fat fraction | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Hepatic iron concentration | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Plasma ghrelin levels | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Adiponectin levels | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Leptin levels | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Blood pressure | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Lipid profile | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Microalbuminuria | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Inflammatory markers (Plasminogen activator inhibitor-1 (PAI-1), C-reactive protein (CRP), homocysteine, tumor necrosis factor (TNF)-α, Interleukin (IL)-6) | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Self-paced step test (Heart rate recovery after exercise) | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Peripheral Arterial Tonometry (PAT) | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Females only: Markers of polycystic ovarian syndrome (PCOS) - Adrenal androgens (17 Hydroxyprogesterone, Dehydroepiandrosterone), sex hormone binding globulin (SHBG), free testosterone, LH/FSH ratio | Baseline (month 0), post 3-month intervention (month 4), and post 6-month extension (month 10).
Females only: Menstrual pattern | Throughout study
Ethnic stratification (Hispanic, African American or Caucasian) | Baseline (month 0)

CONTACTS AND LOCATIONS:
Overall Officials: Tania S Burgert, MD, Principal Investigator — Yale University Medical School
Locations (1):
- Yale Center for Clinical Investigation (YCCI), New Haven, Connecticut, United States

REFERENCES:
- [Result] Burgert TS, Duran EJ, Goldberg-Gell R, Dziura J, Yeckel CW, Katz S, Tamborlane WV, Caprio S. Short-term metabolic and cardiovascular effects of metformin in markedly obese adolescents with normal glucose tolerance. Pediatr Diabetes. 2008 Dec;9(6):567-76. doi: 10.1111/j.1399-5448.2008.00434.x. Epub 2008 Aug 27. PMID 18761646